CLINICAL TRIAL: NCT03437564
Title: A Randomized, Open-Label, 2×2 Crossover Phase 1 Study to Evaluate the Bioequivalence of Single Oral Dose of Lu AA21004 20 mg Tablet and 2× Lu AA21004 10 mg Tablets in Healthy Adult Subjects
Brief Title: A Bioequivalence Study of the Lu AA21004 20 mg and 2×10 mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Vortioxetine-1001; U1111-1208-2715 (Other: WHO); JapicCTI-183863 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Healthy Adult Participants
MeSH Terms: interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vortioxetine one 20 mg tablet + two 10 mg tablets (Experimental): Vortioxetine 20 mg (one 20 mg tablet) on Day 1 in Period 1 in a fasted state + vortioxetine 20 mg (two 10 mg tablets) on Day 1 in Period 2 in a fasted state.
  Interventions: Drug: Vortioxetine
- Vortioxetine two 10 mg tablets + one 20 mg tablet (Experimental): Vortioxetine 20 mg (two 10 mg tablets) on Day 1 in Period 1 in a fasted state + vortioxetine 20 mg (one 20 mg tablet) on Day 1 in Period 2 in a fasted state.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Vortioxetine tablet
  Other Names: Lu AA21004

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of a single oral administration of a vortioxetine (Lu AA21004) 20 mg tablet in comparison with two of vortioxetine 10 mg tablets in Japanese healthy adult participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called vortioxetine (Lu AA21004). Vortioxetine is being tested in Japanese healthy adult participants. This study will look at the bioequivalence of a single oral administration of a vortioxetine 20 mg tablet in comparison with two of vortioxetine 10 mg tablets, and also look at the safety of a single oral dose of vortioxetine 20 mg in Japanese healthy adult participants.

The study will enroll 28 (14 for each sequence) healthy participants. In case bioequivalence cannot be demonstrated with the number of participants initially planned, an add-on participant study may be conducted (as a maximum 28 participants additionally). Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups.

* Treatment Group A: Vortioxetine 20 mg (one 20 mg tablet) in Period 1 + Vortioxetine 20 mg (two 10 mg tablets) in Period 2
* Treatment Group B: Vortioxetine 20 mg (two 10 mg tablets) in Period 1 + Vortioxetine 20 mg (one 20 mg tablet) in Period 2

This single-center trial will be conducted in Japan. The overall time to participate in this study is approximately 25 days. Participants will make two visits to the clinic and be hospitalized for ten days in total.

ELIGIBILITY:
Inclusion Criteria:

1. Be a healthy Japanese adult volunteer.
2. Understand the contents of the study and is capable of providing written consent to participate in the study.
3. Be willing to comply with all study procedures and restrictions.
4. Aged between ≥20 and ≤45 years at the time of screening.
5. Have a BMI of ≥18.5 and ≤24.9 (kg/m^2) and a body weight of ≥50 kg at the time of screening.
6. Be a extensive metabolizer (EM) based on CYP2D6 genotyping at the time of screening.
7. A female participant of childbearing potential with a non-sterilized male partner must agree to routinely use appropriate contraception during the study from the time of signing informed consent until 4 weeks after last dosing of the study drug.

Exclusion Criteria:

1. Has received any investigational drug within 90 days before screening for this study.
2. Previously received Lu AA21004 before participation in this study.
3. Is an employee of the sponsor or the study site, or immediate family member, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or who may be coerced to provide consent.
4. Has uncontrolled, clinically relevant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality which may affect study participation or study results.
5. Has a history of multiple episodes or severe allergies (eg, food, drug, latex allergy) or has had an anaphylactic reaction or significant intolerance to prescription drugs, over the counter (OTC) drugs, or foods.
6. Has a positive pregnancy test at the time of screening or Day -1.
7. Is a pregnant or lactating female.
8. Has a positive urine drug screen test at the time of screening or Day -1.
9. Has a history of drug abuse (defined as any illicit drug use) or has a history of alcohol dependence within 2 years before the start of screening or is unwilling to agree to abstain from alcohol and drugs throughout the study.
10. Consumes 6 or more servings of caffeinated beverages (containing about 120 mg of caffeine per serving) such as of coffee, tea, cola, or energy drinks.
11. Is a smoker who smoked cigarettes or used nicotine-containing products (such as nicotine patch) within 6 months before the Period 1 study drug administration.
12. Used any of the excluded drugs, dietary products or foods during the specified time periods, or will need any of them during the study period.
13. Has any current or recent gastrointestinal diseases that would be expected to influence the absorption of drugs (ie, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn), or any surgical intervention (Stomach, cholecystectomy etc.).
14. Has a history of cancer.
15. Has a positive test result for any of the following at the time of screening: hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody/antigen, serological test for syphilis.
16. Has poor peripheral venous access.
17. Has undergone whole blood collection of at least 200 mL within 4 weeks (28 days) or at least 400 mL within 12 weeks (84 days) prior to the start of Period 1 study drug administration.
18. Has undergone whole blood collection of at least 800 mL in total within 52 weeks (364 days) prior to the start of Period 1 study drug administration.
19. Has undergone blood component collection within 2 weeks (14 days) prior to the start of Period 1 study drug administration.
20. Has any clinically relevant abnormality in vital signs or 12-lead electrocardiograms (ECG) at screening or on Day -1 of Period 1.
21. Has abnormal laboratory test values at screening or on Day -1 of Period 1 indicating clinically relevant underlying disease, or showing alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5×upper limit of normal (ULN).
22. Is unlikely to comply with the protocol requirements or is unsuitable as a participant of this study for any other reason in the opinion of the investigator or sub-investigator.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Nishi Kumamoto Hospital, Kumamoto, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan, from 16 February 2018 to 13 April 2018.
Pre-assignment Details: Healthy participants were enrolled in one of two treatment group (vortioxetine 20 mg (1×20 mg tablet) on Day 1 in Period 1, followed by vortioxetine 20 mg (2×10 mg tablets) on Day 1 in Period 2; vortioxetine 20 mg (2×10 mg tablets) on Day 1 in Period 1, followed by vortioxetine 20 mg (1×20 mg tablet) on Day 1 in Period 2) with cross over design.
Groups:
- Vortioxetine One 20 mg Tablet + Two 10 mg Tablets: Vortioxetine 20 mg (one 20 mg tablet) orally, once on Day 1 in Period 1 in a fasted state + vortioxetine 20 mg (two 10 mg tablets) orally, once on Day 1 in Period 2 in a fasted state.
- Vortioxetine Two 10 mg Tablets + One 20 mg Tablet: Vortioxetine 20 mg (two 10 mg tablets) orally, once on Day 1 in Period 1 in a fasted state + vortioxetine 20 mg (one 20 mg tablet) orally, once on Day 1 in Period 2 in a fasted state.
Period: Overall Study
Arm/Group | Vortioxetine One 20 mg Tablet + Two 10 mg Tablets | Vortioxetine Two 10 mg Tablets + One 20 mg Tablet
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pharmacokinetic (PK) Analysis Set; PK analysis set included all treated participants who had no major protocol violations, completed the minimum element of the protocol, and had evaluable pharmacokinetic data.
Groups:
- Vortioxetine Two 10 mg Tablets + One 20 mg Table: Vortioxetine 20 mg (two 10 mg tablets) orally, once on Day 1 in Period 1 in a fasted state + vortioxetine 20 mg (one 20 mg tablet) orally, once on Day 1 in Period 2 in a fasted state.
- Total: Total of all reporting groups
Arm/Group | Vortioxetine One 20 mg Tablet + Two 10 mg Tablets | Vortioxetine Two 10 mg Tablets + One 20 mg Table | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.0 (6.52) | 24.0 (4.96) | 24.0 (5.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 14 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 14 | 14 | 28
Height [Mean (Standard Deviation); unit: Centimeters (cm)] | 172.4 (3.94) | 170.2 (6.48) | 171.3 (5.38)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 63.86 (6.694) | 61.91 (6.254) | 62.89 (6.434)
BMI [Mean (Standard Deviation); unit: kg/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/meter (m)^2 | 21.46 (1.812) | 21.33 (1.175) | 21.39 (1.500)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 12 | 13 | 25
  Ex-Smoker | 2 | 1 | 3
Alcohol Classification [Count of Participants; unit: Participants]
  Drank 2 to 3 Days a Week | 3 | 0 | 3
  Drank 2 to 3 Days a Month | 9 | 8 | 17
  Never Drank | 2 | 6 | 8
Caffeine Classification [Count of Participants; unit: Participants]
  Had Caffeine Consumption | 5 | 4 | 9
  Had no Caffeine Consumption | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Last Quantifiable Time Point of Unchanged Lu AA21004
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- Vortioxetine One 20 mg Tablet: Vortioxetine 20 mg (one 20 mg tablet) orally, once on Day 1 in Period 1 in a fasted state plus Day 1 in Period 2 in a fasted state.
- Vortioxetine Two 10 mg Tablets: Vortioxetine 20 mg (two 10 mg tablets) orally, once on Day 1 in Period 1 in a fasted state plus Day 1 in Period 2 in a fasted state.
Arm/Group | Vortioxetine One 20 mg Tablet | Vortioxetine Two 10 mg Tablets
Number analyzed (Participants) | 28 | 28
hour*nanogram per milliliter (h*ng/mL) | 299.3 (59.820) | 301.1 (62.070)
Statistical Analysis 1: Comparison: Vortioxetine One 20 mg Tablet vs Vortioxetine Two 10 mg Tablets; Test type: Equivalence — The difference in the least square (LS) means between the formulations (dosing of one Vortioxetine 20 mg tablet - dosing of two Vortioxetine 10 mg tablets) and the two-sided 90% confidence interval (CI) were provided using a crossover analysis of variance (ANOVA) model. The shown data were anti-logs of LS means difference and CI. The ANOVA model included log-transformed (natural log) PK parameters AUClast as dependent variable, and treatment condition, group, and period as independent variables; ANOVA; Point Estimate = 0.996, 90% CI 2-sided [0.967 to 1.026]

2. Primary Outcome: Cmax: Maximum Plasma Concentration (Observed Value) of Unchanged Lu AA21004
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vortioxetine One 20 mg Tablet | Vortioxetine Two 10 mg Tablets
Number analyzed (Participants) | 28 | 28
ng/mL | 8.744 (1.7838) | 8.976 (1.6936)
Statistical Analysis 1: Comparison: Vortioxetine One 20 mg Tablet vs Vortioxetine Two 10 mg Tablets; Test type: Equivalence — The difference in the LS means between the formulations (dosing of one vortioxetine 20 mg tablet - dosing of two vortioxetine 10 mg tablets) and the two-sided 90% CI were provided using a crossover ANOVA model. The shown data were anti-logs of LS means difference and CI. The ANOVA model included log-transformed (natural log) PK parameters Cmax as dependent variable, and treatment condition, group, and period as independent variables; ANOVA; Point Estimate = 0.972, 90% CI 2-sided [0.937 to 1.008]

3. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity of Unchanged Lu AA21004
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Vortioxetine One 20 mg Tablet | Vortioxetine Two 10 mg Tablets
Number analyzed (Participants) | 28 | 28
h*ng/mL | 463.9 (135.58) | 477.6 (164.83)

4. Secondary Outcome: Tmax: Time to Reach Cmax (Observed Value) of Unchanged Lu AA21004
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Hours
Arm/Group | Vortioxetine One 20 mg Tablet | Vortioxetine Two 10 mg Tablets
Number analyzed (Participants) | 28 | 28
Hours | 6.000 [6.00 to 8.00] | 6.000 [6.00 to 8.00]

5. Secondary Outcome: MRT∞, ev: Mean Residence Time 0 to Infinity of Unchanged Lu AA21004
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Vortioxetine One 20 mg Tablet | Vortioxetine Two 10 mg Tablets
Number analyzed (Participants) | 28 | 28
Hours | 67.27 (14.145) | 68.84 (18.646)

6. Secondary Outcome: MRTlast, ev: Mean Residence Time From Time 0 to the Time of the Last Quantifiable Concentration of Unchanged Lu AA21004
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Vortioxetine One 20 mg Tablet | Vortioxetine Two 10 mg Tablets
Number analyzed (Participants) | 28 | 28
Hours | 30.12 (1.8274) | 30.12 (1.8335)

7. Secondary Outcome: λz: Apparent Elimination Rate Constant of Unchanged Lu AA21004
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: 1/Hours
Arm/Group | Vortioxetine One 20 mg Tablet | Vortioxetine Two 10 mg Tablets
Number analyzed (Participants) | 28 | 28
1/Hours | 0.01608 (0.0040090) | 0.01599 (0.0041766)

8. Secondary Outcome: T1/2z: Apparent Elimination Half-Life of Unchanged Lu AA21004
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Vortioxetine One 20 mg Tablet | Vortioxetine Two 10 mg Tablets
Number analyzed (Participants) | 28 | 28
Hours | 45.36 (9.7694) | 46.44 (13.090)

9. Secondary Outcome: Number of Participants Who Experienced at Least One Treatment-Emergent Adverse Event (TEAE)
Time Frame: Up to Day 25
Population: Safety Analysis Set; The safety analysis set included all participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Vortioxetine One 20 mg Tablet | Vortioxetine Two 10 mg Tablets
Number analyzed (Participants) | 28 | 28
Participants | 1 | 0

10. Secondary Outcome: Number of Participants With TEAE Related to Vital Sign
Time Frame: Up to Day 25
Population: Safety Analysis Set; The safety analysis set included all participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Vortioxetine One 20 mg Tablet | Vortioxetine Two 10 mg Tablets
Number analyzed (Participants) | 28 | 28
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With TEAE Related to Clinical Laboratory Tests (Alanine Aminotransferase Increased)
Time Frame: Up to Day 25
Population: Safety Analysis Set; The safety analysis set included all participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Vortioxetine One 20 mg Tablet | Vortioxetine Two 10 mg Tablets
Number analyzed (Participants) | 28 | 28
Participants | 1 | 0

12. Secondary Outcome: Number of Participants With TEAE Related to 12-lead Electrocardiograms
Time Frame: Up to Day 25
Population: Safety Analysis Set; The safety analysis set included all participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Vortioxetine One 20 mg Tablet | Vortioxetine Two 10 mg Tablets
Number analyzed (Participants) | 28 | 28
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 25
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Vortioxetine One 20 mg Tablet | Vortioxetine Two 10 mg Tablets
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 1/28 | 0/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine One 20 mg Tablet (N=28) | Vortioxetine Two 10 mg Tablets (N=28)
Alanine aminotransferase increased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT03437564/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT03437564/SAP_001.pdf